CLINICAL TRIAL: NCT03285529
Title: The Use of STRATAFIX Suture Device Compared to Standard-of-care for Deep Tissue Closure in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Viktor Krebs, M.D., Vice Chairman - Adult Reconstruction, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-841
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Wound; Knee
Keywords: barbed suture; knoteless suture; total knee arthroplasty; wound; closure; time
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- STRATAFIX GROUP (Active Comparator): STRATIFIX symmetric PDS Plus #1 will be used to close the capsule following total knee arthroplasty. The subcutaneous layer will be then closed with simple interrupted knots using number 2-0 braided absorbable sutures (Vicryl), followed by closure of the subcutaneous layer using a number 2-0 monofilament absorbable suture with inverted interrupted knots (Monocryl) followed by the use of steri-strips and adhesive
  Interventions: Device: STRATIFIX
- CONTROL GROUP (Placebo Comparator): The arthrotomy (deep layer) is repaired using Vicryl #1 followed by closure of the intermediate layer with a 2-0 Vicryl and a subcutaneous layer with a 2-0 Monocryl followed by steri-strips and adhesive, following total knee arthroplasty.
  Interventions: Device: VICRYL

INTERVENTIONS:
Device: STRATIFIX — STRATIFIX symmetric PDS Plus; Stratifix knotless suture
  Arms: STRATAFIX GROUP
Device: VICRYL — Vicryl #1
  Arms: CONTROL GROUP

SUMMARY:
The STRATAFIX (Ethicon, Johnson and Johnson, Somerville, New Jersey) Knotless Tissue Control suture device is a barbed suture that uses anchor technology to securely engage with the soft tissues while also eliminating the need for knots. The anchors, or barbs, are pressed out of the device core or formed within the core in a geometric pattern and arranged in a tapered manner to allow the device to pass through tissue in the direction toward the needle during closure. These knotless tissue control devices are deployed using a continuous technique, which is anticipated to be faster and more cost-effective than interrupted suturing.

DETAILED DESCRIPTION:
Preclinical and biomechanical studies have demonstrated efficacy in cosmetic skin and deep tissue closures.[1], [2] In addition, barbed sutures have been shown to provide water-tight closure and wound strength comparable to or superior to closure with conventional sutures. Many comparative studies have been published contrasting barbed sutures to conventional closure techniques in multiple surgical fields. [3], [4] Various studies have evaluated the outcomes of different barbed suture devices, however there are no reports assessing the length of closure times using STRATAFIX (Ethicon, Johnson and Johnson, Somerville, New Jersey) Knotless Tissue Control Devices during deep closure in total hip arthroplasty. Stephens et al. [5] performed a prospective randomized study of 500 total knee arthroplasty patients who received either barbed suture (250) or conventional sutures (250) for deep closure of the surgical wound. The mean operating time was significantly shorter in the barbed group as compared to conventional group (64.3 vs 68.1 minutes, p=<0.001). In a study of 80 TKA (61 barbed, 19 conventional deep sutures) and 54 THA patients (37 barbed, 17 conventional deep sutures), Smith et al. [6] found significantly shorter closure time in the barbed suture group (16.78 vs. 26.5 minutes, p<0.001). One study reports one the use of Stratfix suture for intracorporeal suturing in myomectomy. Giampaolino et al. [7] performed a prospective randomized study on 47 patients and evaluated the mean operative time for laparoscopic posterior myomectomy using Stratafix or conventional suture for intracorporeal suturing. There was a significant decrease in mean operative time associated with use of Stratafix suture as compared to conventional suture (66.3 vs 73 minutes, p=0.005).

This prospective randomized single-center study will examine the outcomes, mainly closure time, of deep closure during total knee arthroplasty using the STRATAFIX Symmetric PDS Plus (Ethicon, Johnson and Johnson, Somerville, New Jersey) barbed suture compared to interrupted VICRYL suture (Ethicon, Johnson and Johnson, Somerville, New Jersey).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, between the ages of 18 to 80 years at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Able to fluently speak and understand the local language
5. If female, is non-pregnant (negative pregnancy test results at the baseline/randomization visit) and non-lactating.
6. End-stage osteoarthritis patients planning to undergo primary total knee arthroplasty
7. BMI less than 40 kg/m2

Exclusion Criteria:

1. BMI greater than or equal to 40 kg/m2.
2. History of known bleeding disorder.
3. History of medical co-morbidity that may result in poor wound healing (i.e. diabetes mellitus, peripheral vascular disease).
4. Patients <18 or >80 years of age.
5. Patients who are prisoners.
6. Mentally unable to sign informed consent.
7. Has an uncontrolled illness that, in the opinion of the investigator, is likely to cause the patient to be withdrawn from the trial or would otherwise interfere with interpreting the results of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Krebs, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.

REFERENCES:
- [Derived] Sundaram K, Warren JA, Klika A, Piuzzi NS, Mont MA, Krebs V. Barbed sutures reduce arthrotomy closure duration compared to interrupted conventional sutures for total knee arthroplasty: a randomized controlled trial. Musculoskelet Surg. 2021 Dec;105(3):275-281. doi: 10.1007/s12306-020-00654-y. Epub 2020 Mar 7. PMID 32146687

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STRATAFIX GROUP | CONTROL GROUP
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: total knee arthroplasty patients
Groups:
- Total: Total of all reporting groups
Arm/Group | STRATAFIX GROUP | CONTROL GROUP | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (7) | 66 (7) | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 14 | 13 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Wound length [Mean (Standard Deviation); unit: centimeters] | 17.1 (2.0) | 16.1 (1.3) | 16.6 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Time to Close, Minutes
Description: Time from first needle insertion to complete skin closure per protocol
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | STRATAFIX GROUP | CONTROL GROUP
Number analyzed (Participants) | 30 | 30
minutes | 19 (0.08) | 28 (0.13)

2. Secondary Outcome: Number of Participants With Wound Complications
Description: superficial wound infection, deep wound infection, periprosthetic joint infection, wound hematoma, and wound dehiscence.
Time Frame: 90 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | STRATAFIX GROUP | CONTROL GROUP
Number analyzed (Participants) | 30 | 30
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 90 days postoperative
Arm/Group | STRATAFIX GROUP | CONTROL GROUP
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STRATAFIX GROUP (N=30) | CONTROL GROUP (N=30)
Superficial surgical site infection (Infections and infestations) | 1 | 0
Wound dehiscence (Infections and infestations) | 0 | 1
Wound hematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
Stitch abscess (Infections and infestations) | 1 | 0
Wound discharge (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03285529/Prot_SAP_001.pdf